CLINICAL TRIAL: NCT07104695
Title: Studying the Feasibility and Acceptability of the SOLOMIYA App - a Smartphone-Based Intervention for People Living Under Prolonged Stress Due to the Ongoing War in Ukraine
Brief Title: Solomiya App - CBT-based Self-help Intervention
Acronym: SOLOAPP-FAIT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Solveig Kemna (Other)
Collaborators: Bogomolets National Medical University (Other)
Responsible Party: Sponsor-Investigator, Solveig Kemna, Dr. med., Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SOL2025UA-DIGIINTV-001
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Stress - Prevention of Sleep Disorders, PTSD and Depression
Keywords: Mobile intervention; Chronic stress; Feasibility
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Solomiya App - CBT-based self-help intervention (Experimental): The Solomiya app is a mobile-based self-help intervention designed to reduce and cope with depressive symptoms and improve sleep in individuals exposed to chronic stress. It has been created within the Solomiya project and is based on preliminary work in other international health settings (Böge 2022) where it has shown to improve depressive symptoms as part of a Stepped Care and Collaborative Model (SCCM). It includes psychoeducational multimedia modules on stress management and sleep problems, along with cognitive behavioral therapy (CBT)-based tools such as guided relaxation exercises, mindfulness practices, and behavioral activation strategies. The app also offers symptom tracking using the PHQ-9 to support user self-monitoring. Participants are instructed to engage with the app regularly over a 4 week period. The intervention is entirely self-guided and does not involve therapist support. App usage and adherence data will be collec
  Interventions: Behavioral: Solomiya App - CBT-based self-help intervention

INTERVENTIONS:
Behavioral: Solomiya App - CBT-based self-help intervention — Solomiya App - CBT-based self-help intervention
  The Solomiya app is a mobile-based self-help intervention designed to reduce and cope with depressive symptoms and improve sleep in individuals exposed to chronic stress. It has been created within the Solomiya project and is based on preliminary work in other international health settings (Böge 2022) where it has shown to improve depressive symptoms as part of a Stepped Care and Collaborative Model (SCCM). It includes psychoeducational multimedia modules on stress management and sleep problems, along with cognitive behavioral therapy (CBT)-based tools such as guided relaxation exercises, mindfulness practices, and behavioral activation strategies. The app also offers symptom tracking using the PHQ-9 to support user self-monitoring. Participants are instructed to engage with the app regularly over a 4 week period. The intervention is entirely self-guided and does not involve therapist support. App usage and adherence data will be collect

SUMMARY:
The project aims to investigate the feasibility and acceptability of a smartphone intervention for depressive symptoms and insomnia in people living under prolonged stress due to the ongoing war in Ukraine. A secondary aim is to assess the clinical outcomes of the intervention by comparing changes in symptoms from baseline (T0) to post-intervention (T1) (single-arm feasibility design). The participants will receive an app-based smartphone intervention with psychoeducational content, relaxation exercises and mindfulness-based interventions and symptom tracking.

DETAILED DESCRIPTION:
Participants will be recruited via Educational - scientific institute of mental health of the Bogomolets National Medical University. An online eligibility screening will be conducted prior to study inclusion via a secure form.

The SOLOMIYA app has been created within the Solomiya project (available on iOS (App Store) and Android (Google Play) platforms) and is based on preliminary work in other international health settings (Böge 2022). It combines psychoeducational multimedia content (e.g., on stress management and sleep problems) and evidence-based CBT-based therapy tools such as relaxation and mindfulness techniques. The app enables users to self-monitor stress symptoms using the PHQ-9 scale.

Participants will carry out self-reported assessments at baseline (T0) and after the intervention phase of 4-6 weeks (T1). App feasibility and acceptability will be evaluated via user behaviour, particularly in terms of adoption, retention and dropout.

User behaviour data will be collected via aggregated app usage metrics as well as user-approved in-app tracking of individual usage patterns, including session frequency and engagement with specific features. Mental health parameters such as depressive symptoms, psychological distress, and sleep quality will be assessed using standardised, validated questionnaires administered at T0 and T1.

The data management plan includes standard procedures for data-handling such as using anonymized identification codes for patient data. The data will be collected and saved in a GDPR-compliant online database (REDCap) on German servers, only allowing researchers involved in the study to access the data.

ELIGIBILITY:
Inclusion Criteria:

* Civilians
* Be in possession of a smartphone
* Be minimum 18 years of age
* Sufficient knowledge of Ukrainian or Russian
* Mild or moderate depression or distress (PHQ-9 score 5-14) OR mild or moderate insomnia symptoms (ISI score 8-21)

Exclusion Criteria:

* Acute suicidal tendencies (defined as a score of 1 or greater on item 9 of the PHQ-9)
* Moderately severe depression (defined as a PHQ-9 score of 15 or more)
* Severe insomnia (defined as a ISI score of 22 or more)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Solomiya app | Post-intervention (4 weeks from baseline)
  Feasibility will be assessed using predefined progression criteria concerning
  * Adoption (initial uptake/ download rates/ completion of onboarding)
  * Retention rates measured by completion of the app modules
  * Rate of participants considered as having dropped out Feasibility will be assessed using predefined progression criteria based on recruitment, engagement, retention, and safety, which are detailed below. The criteria will be operationalized with an approach using traffic-light benchmarks (Avery 2017).
Acceptability of Solomiya app | Post-intervention (4 weeks from baseline)
  Acceptability will be assessed by using the Client Satisfaction Questionnaire (Attkisson & Zwick, 1982) and a series of open-ended questions about app usability, relevance and acceptability. No serious adverse events related to app use are expected.

SECONDARY OUTCOMES:
Depressive Symptoms | At baseline and post-intervention (4 weeks from baseline)
  Patient Health Questionnaire - 9 (Kroenke, 2001). The Patient Health Questionnaire-9 (PHQ-9) is a 9-item scale assessing depressive symptoms (Kroenke et al., 2001). Scores range from 0 to 27, with higher scores indicating worse outcomes (i.e., more severe depression).
Sleep quality | At baseline and post-intervention (4 weeks from baseline)
  Insomnia Severity Index (ISI) (Bastien 2001). The Insomnia Severity Index (ISI) is a 7-item scale measuring the nature, severity, and impact of insomnia (Bastien et al., 2001). Scores range from 0 to 28, with higher scores indicating worse outcomes, i.e., more severe insomnia.
Resilience | At baseline and post-intervention (4 weeks from baseline). The Brief Resilience Scale (BRS) is a 6-item scale designed to assess the ability to recover from stress (Smith et al., 2009). Scores range from 1 to 5, averaged across items, with higher scores
  Brief Resilience Scale (Smith 2009)

CONTACTS AND LOCATIONS:
Locations (1):
- Bogomolets National Medical University, Kyiv, Kyiv Oblast, Ukraine

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Smith BW, Dalen J, Wiggins K, Tooley E, Christopher P, Bernard J. The brief resilience scale: assessing the ability to bounce back. Int J Behav Med. 2008;15(3):194-200. doi: 10.1080/10705500802222972. PMID 18696313
- [Background] Boge K, Karnouk C, Hoell A, Tschorn M, Kamp-Becker I, Padberg F, Ubleis A, Hasan A, Falkai P, Salize HJ, Meyer-Lindenberg A, Banaschewski T, Schneider F, Habel U, Plener P, Hahn E, Wiechers M, Strupf M, Jobst A, Millenet S, Hoehne E, Sukale T, Dinauer R, Schuster M, Mehran N, Kaiser F, Brocheler S, Lieb K, Heinz A, Rapp M, Bajbouj M. Effectiveness and cost-effectiveness for the treatment of depressive symptoms in refugees and asylum seekers: A multi-centred randomized controlled trial. Lancet Reg Health Eur. 2022 Jun 6;19:100413. doi: 10.1016/j.lanepe.2022.100413. eCollection 2022 Aug. PMID 35694653
- [Background] Avery KN, Williamson PR, Gamble C, O'Connell Francischetto E, Metcalfe C, Davidson P, Williams H, Blazeby JM; members of the Internal Pilot Trials Workshop supported by the Hubs for Trials Methodology Research. Informing efficient randomised controlled trials: exploration of challenges in developing progression criteria for internal pilot studies. BMJ Open. 2017 Feb 17;7(2):e013537. doi: 10.1136/bmjopen-2016-013537. PMID 28213598